CLINICAL TRIAL: NCT06649903
Title: Comparison of Cervical Spinal Manipulation and Visceral Osteopathy Techniques in People with Mechanical Neck Pain
Brief Title: Cervical Spinal Manipulation and Visteral Osteopathy for Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Hilal Denizoğlu Külli, Assoc. Prof., Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cihat Seyrek
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Neck Pain
Keywords: neck pain treatment; visceral osteopathy; servical spinal manupilation; osteopathy
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Chiropractic; Osteopathic Physicians

STUDY DESIGN:
Intervention Model Description: It is a randomized controlled study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cervical Spinal Manipulation (CSM) (Experimental): This arm includes participants who receive a single session of high-velocity, low-amplitude spinal manipulation aimed at reducing pain and improving cervical range of motion and muscle strength in individuals with mechanical neck pain. The intervention is administered by a qualified physiotherapist, following established protocols for cervical spinal manipulation.
  Interventions: Behavioral: Chiropractic
- Visceral Osteopathy (Experimental): Participants in this arm undergo a single session of visceral osteopathy techniques focused on improving pain and functional outcomes in individuals with mechanical neck pain. The VO techniques are designed to enhance mobility and alleviate discomfort through manipulation of the viscera and associated structures, performed by a trained osteopath.
  Interventions: Behavioral: Osteopathy

INTERVENTIONS:
Behavioral: Chiropractic — high speed low amplitude neck manipulation
  Arms: Cervical Spinal Manipulation (CSM)
Behavioral: Osteopathy — the stomach and liver technique was applied
  Arms: Visceral Osteopathy

SUMMARY:
This study compares two treatment techniques, cervical spinal manipulation (CSM) and visceral osteopathy (VO), in patients with mechanical neck pain (MNP). The aim of the study was to evaluate the effects of these treatments on pain levels, neck mobility, and muscle strength in both the neck and upper extremities.

DETAILED DESCRIPTION:
The purpose of this study is to compare the acute effects of cervical spinal manipulation (CSM) treatment and visceral osteopathy (VO) techniques on pain, cervical range of motion (ROM), muscle strength, and grip strength in individuals with mechanical neck pain (MNP).

The study is going to include a total of 30 subjects aged 18-60 diagnosed with MNP. The subjects are randomly divided into two groups. The CSM group received high-velocity, low-amplitude (HVLA) spinal manipulation, while the other group underwent VO techniques. Each treatment technique is going to be applied in only one session. Pain intensity is assessed using the Visual Analog Scale (VAS). Cervical ROM and the craniovertebral angle (CVA) are evaluated using a goniometer. Neck and elbow muscle strength are measured with a hand-held dynamometer, and grip strength is assessed using a hand-grip dynamometer.

ELIGIBILITY:
Inclusion Criteria:

* Participants is included if they had neck pain present for at least one week, reduced cervical ROM, a manual muscle test score of 4 or higher for the neck muscles, and no neurological pain in the neck.

Exclusion Criteria:

* Exclusion criteria included individuals with rheumatic diseases, a history of spinal surgery, neck fractures, tumors in the neck region, vertebrobasilar artery insufficiency, blood clotting disorders, or inadequate mental capacity.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
VAS pain scale | At baseline and immediately following the intervention session.
  The Visual Analog Scale (VAS) for pain is a subjective measurement tool used to assess an individual's pain intensity. It consists of a straight line, typically 10 centimeters in length, with endpoints that represent the extremes of pain: one end signifies "no pain" (0) and the other indicates "worst pain imaginable" (10).
  Participants mark a point on the line that corresponds to their pain level at the moment of assessment. The distance from the "no pain" end to the marked point is then measured in centimeters, providing a numerical value that quantifies the intensity of the pain experienced. This scale is commonly used in clinical settings for its simplicity and effectiveness in capturing the subjective experience of pain.
Microfet 2 Dynamometer | At baseline and immediately following the intervention session.
  The Microfet 2 Dynamometer is a handheld device used to objectively measure muscle strength in clinical and research settings. It employs a digital force transducer that provides accurate and reliable assessments of isometric muscle strength across various muscle groups.
  It is commonly used in physical therapy and rehabilitation to evaluate muscle function, track progress over time, and inform treatment decisions. Its compact size and versatility make it suitable for various assessments, including grip strength, limb strength, and specific muscle testing. The device is particularly valuable for ensuring standardized measurements in strength evaluation protocols.

SECONDARY OUTCOMES:
Hand Dynamometer | At baseline and immediately following the intervention session.
  A hand dynamometer is a electronic device used to measure grip strength, which is an important indicator of overall muscle strength and function.
  The hand dynamometer is widely used in clinical, rehabilitation, and research settings to assess the strength of the hand and forearm muscles. This measurement can provide valuable information regarding a patient's recovery progress, functional capacity, and overall health status.
  Consistent use of the hand dynamometer can help establish baselines, track changes in muscle strength over time, and guide treatment interventions for various conditions affecting hand function.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Atlas University, Istanbul, Kagıthane
  - Atlas University, Istanbul, Kağıthane

IPD SHARING:
Plan to Share IPD: No
At this time, we are undecided about sharing individual participant data (IPD) with other researchers. We will evaluate the feasibility and ethical considerations of data sharing upon study completion. Factors influencing this decision may include participant confidentiality, data integrity, and potential research collaborations. A final determination will be made based on these considerations to ensure compliance with ethical guidelines and the responsible use of participant data.